CLINICAL TRIAL: NCT02236481
Title: No-profit" Study to Ensure Normal Clinical Practice, to Evaluate the Efficacy of Anakinra in Reducing the Glycated Haemoglobin in Patients Affected by Rheumatoid Arthritis and Diabetes; Randomized, Open Label, Parallel Group,Controlled Clinical Study
Brief Title: Clinical Study to Evaluate the Efficacy of Anakinra in Patients With Rheumatoid Arthritis and Diabetes
Acronym: TRACK
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Decision of the Sponsor for Early Benefits
Sponsor: Prof. Roberto Giacomelli (Other)
Responsible Party: Sponsor-Investigator, Prof. Roberto Giacomelli, Full Professor of Rheumatology, University of L'Aquila
Organization: University of L'Aquila (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRACK
Record Dates: First submitted 2014-09-08; First posted 2014-09-10 (Estimated); Last update posted 2018-12-14 (Actual); Status verified 2018-12

CONDITIONS: Diabetes Mellitus, Type 2; Arthritis, Rheumatoid
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Arthritis, Rheumatoid | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anakinra (Experimental): 100 mg of anakinra once daily by subcutaneous injection for 24 months
  Interventions: Drug: Anakinra
- TNF alpha inhibitors (Active Comparator): treatment with TNF-alpha inhibitors according to the relative summary of product charateristics
  Interventions: Drug: TNF alpha inhibitors

INTERVENTIONS:
Drug: Anakinra
  Other Names: Kineret
  Arms: Anakinra
Drug: TNF alpha inhibitors
  Arms: TNF alpha inhibitors

SUMMARY:
The TRACK [Treatment of Rheumatoid Arthritis and Comorbidities with Kineret (anakinra)]-study: a randomized, open-label multicenter study assessing the efficacy of anakinra in lowering HbA1c (glycated hemoglobin) as well as changes in DAS28 in Rheumatoid Arthritis (R.A.) patients with type 2 diabetes (T2D) Authors: R. Giacomelli,(A,B) P. Cipriani (A) and P. Ruscitti (A) on behalf of the TRACK study-group; (A) University of L'Aquila, L'Aquila, Italy; Background: Interleukin-1 (IL-1) plays a pivotal role in R.A., joint erosion and cartilage destruction.(1) Anakinra (a recombinant form of the naturally occurring IL-1 receptor antagonist (IL-1Ra), which blocks the activity of both IL-1α and IL-1β) has shown in a number of RCTs (2-6) to be effective in the treatment of R.A., in monotherapy,(2,4) as well as associated to methotrexate (MTX).(3,5,6) IL-1β plays also an important role in the pathogenesis of T2D: Glucose has been shown to induce IL-1β hypersecretion through inflammasome activation, while IL-1β induces impairment of β-cell secretory function and β-cell apoptosis.(7) In prediabetic subjects, the expression of IL-1Ra is induced by IL-1β and reflects the body's response to counterbalance increased IL-1β activity.(7) Levels of IL-1Ra tend to rise up to 6 years before the diagnosis of T2D.(8,9) IL-1Ra has been successfully used as a marker for the risk of developing T2D in subjects with metabolic syndrome.(10) As a clinical proof of concept, IL-1 inhibition with anakinra in patients with T2D has shown to improve the secretorial function of beta-cells as well as to lower the ratio of proinsulin/insulin and glycated hemoglobin/hemoglobin significantly, favoring glycemic control and possibly reducing the severity and prevalence of the associated complications of this disease.(11) Summarizing, IL-1 inhibition with anakinra has a clinical impact on R.A. as well as T2D. As from 6-10% of Italian R.A. patients have also T2D, this trial aims at investigating the impact of IL-1 inhibition on both diseases. Very recent data also show that T2D is a predictor of response to anakinra-treatment in R.A. patients,(12) which furthermore justifies the use of anakinra in this subset of R.A. patients. Objectives: [Primary] To evaluate the change in HbA1c between baseline, 3 months, 6 months, 1 year and at last follow up of 2 years from the beginning; [Secondary] To evaluate the efficacy on controlling signs & symptoms of R.A., assessing the remission rate at 3 months, 6 months, 1 year and at follow up (2 years), using the evaluation scale of disease activity on 28 joints, DAS28 and SDAI improvements from baseline conditions over time points, according to EULAR response criteria. Methods: 200 patients in 28 Italian centers with active R.A. refractory to treatment with methotrexate and T2D will be enrolled and randomized to receive either 100mg of anakinra once daily by subcutaneous injection or any anti-TNF-alfa drug treatment. [84 subjects will be required in each treatment arm to reach 90% power with an alpha error of 0.05 to detect a mean difference between the study arms of 0.25 percentage points of HbA1c . The assumed difference of HbA1c is rather conservative when compared to previously published changes in T2D patients (11).] Anti-diabetic treatment is required to be unchanged for at least one month prior to enrolment. Patients will be invited to maintain dietary habits and lifestyle during the study period. Further details can be viewed on the trials website after subscription.(13) References: (1) Arend & Dayer, Adv. Imm. 1993; 54: 167-227. (2) Bresnihan, Arthritis Rheum. 1998; 41: 2196-2204. (3) Cohen, Arthritis Rheum. 2002; 46: 614-624. (4) Nuki, Arthritis. Rheum. 2002; 46: 2838-2846. (5) Cohen, ARD 2004; 63: 1062-1068. (6) Cohen, Rheumatology 2004; 43: 704-711. (7) Donath, Nat. Rev. Immunol. 2011; 11: 98-107. (8) Herder, Diabetes Care 2009; 32: 421-423. (9) Carstensen, Diabetes 2010; 59: 1222-1227. (10) Luotola, J. Intern. Med. 2011; 269: 322-332. (11) Larsen, NEJM 2007; 356: 1517-1526. (12) Missler-Karger, EULAR 2013, Abs. FRI0219. (13) http://www.anakinra-ra-diabetes.org/ Disclosure: This trial is receiving support from Swedish Orphan Biovitrum AB according to the Italian law decree 17 December 2004. (B) speaker fees

ELIGIBILITY:
Inclusion Criteria:

* male and female patients aged ≥ 18 years;
* previous diagnosis of RA with criteria of the American College of Rheumatology (ACR) / European League Against Rheumatism (EULAR);
* Diagnosis of Diabetes Mellitus type II according to the American Diabetes Association (ADA) criteria since at least 6 months;
* Patients with an inadequate response to previous treatment with methotrexate (determined on the basis of the evaluation of the physician);
* BMI <35
* Glycated hemoglobin > 7% <10%
* Minimum score Disease Activity Score-28 (DAS 28) > 3.2
* For patients previously treated with a biologic drug, wash out of the treatment for at least 1 month prior to enrollment;
* For patients in treatment with hypoglycemic drugs at enrollment, no change of the hypoglycemic treatment in terms of type of drug and dosage, for a period of at least 3 months before enrolment
* For patients in therapy with other drugs at baseline, no change in terms of drug administered and the dosage regimen for a period of at least 1 month prior to enrollment;
* Absence of signs and symptoms related to ischemic heart disease
* Signature of written Informed Consent Form.

Exclusion Criteria:

* DM2 diagnosed since more than 10 years;
* Ongoing Acute infection or chronic infection, which has one or more of following:

  * Increased levels of C-reactive protein > 30 mg / L
  * fever
  * Ongoing treatment with antibiotics ;
* Chronic granulomatous infections (ie. tuberculosis diagnosed by radiography or by laboratory tests)
* History of recurrent infections or presence of diseases that induce to infections;
* C-peptide values <0.5 ng / mL ( 0.1665 nmol / L)
* presence of neutropenia ( WBC < 2000/mm3 ) or anemia (hemoglobin < 11g/dL for man and 10g/dl for the woman) ;
* presence of one or more contraindication indicate in SmPC of study drug (anakinra);
* presence of one or more contraindication indicate in SmPC of control drug (inhibitors of TNF -alpha ; ATC L04AB);
* presence of one or more contraindications to treatment with methotrexate ;
* previous ischemic attack or myocardial infarction;
* heart failure NYHA class III or IV;
* hepatic or progressive liver disease ( values of ALAT / ASAT increased by at least two -fold compared to normal limits );
* pregnant, or women not using contraceptive measures;
* breast-feeding;
* participation in another clinical study up to 6 months before randomization;
* depressive syndrome or other serious psychiatric illness that, in the opinion of the physician, may preclude participation in the study;
* presence of known malignancy ;
* Clinically significant history of alcohol abuse or drug addiction , that, in the opinion of the physician, may preclude participation in the study;
* any condition that, in the opinion of the physician, precludes the possibility of using the study drug (anakinra , Kineret ) or the control drug (inhibitors of TNF alpha; L04AB ATC ) in compliance with SmPC indications ;
* any other condition or laboratory parameter that , in the opinion of the physician, precludes the subject's participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2013-07; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Glycated Hemoglobin | up to 24th months of treatment

SECONDARY OUTCOMES:
Percentage of patients in remission ( EULAR Criteria ) | baseline , after 3 months, 6 months , 12 months and 24 months of treatment
Percentage of patients improved ( EULAR criteria) | baseline , after 3 months, 6 months , 12 months and 24 months of treatment
Count of tender joints (66 joints) | baseline , after 3 months, 6 months , 12 months and 24 months of treatment
Count of swollen joints (68 joints) | baseline , after 3 months, 6 months , 12 months and 24 months of treatment
Administration at Health Assessment Questionnaire ( HAQ) | baseline , after 3 months, 6 months , 12 months and 24 months of treatment
C-reactive protein (CRP) and erythrocyte sedimentation rate ( ESR ) | baseline , after 3 months, 6 months , 12 months and 24 months of treatment:
Plasma levels of glucose | baseline , after 3 months, 6 months , 12 months and 24 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Giacomelli, Professor, Principal Investigator — University of L'Aquila
Locations (1):
- L'Aquila University, L’Aquila, Italy

REFERENCES:
- [Derived] Ruscitti P, Masedu F, Alvaro S, Airo P, Battafarano N, Cantarini L, Cantatore FP, Carlino G, D'Abrosca V, Frassi M, Frediani B, Iacono D, Liakouli V, Maggio R, Mule R, Pantano I, Prevete I, Sinigaglia L, Valenti M, Viapiana O, Cipriani P, Giacomelli R. Anti-interleukin-1 treatment in patients with rheumatoid arthritis and type 2 diabetes (TRACK): A multicentre, open-label, randomised controlled trial. PLoS Med. 2019 Sep 12;16(9):e1002901. doi: 10.1371/journal.pmed.1002901. eCollection 2019 Sep. PMID 31513665

DOCUMENTS (2):
  • Study Protocol (2012-11-15): https://cdn.clinicaltrials.gov/large-docs/81/NCT02236481/Prot_000.pdf
  • Informed Consent Form (2012-11-15): https://cdn.clinicaltrials.gov/large-docs/81/NCT02236481/ICF_001.pdf